CLINICAL TRIAL: NCT06748937
Title: A Phase 2 Randomized, Open-label Trial to Evaluate the Early Bactericidal Activity, Safety, Tolerability, and Dose-Response of Oral Alpibectir in Combination With Ethionamide, and With Ethionamide, Rifampicin, Pyrazinamide, and Ethambutol in Adults With Newly Diagnosed, Drug-Susceptible Pulmonary Tuberculosis
Brief Title: A Study of the Early Effects, Safety, and Acceptability of Oral Alpibectir in Combination With Ethionamide
Acronym: ENABLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TASK; UNITE4TB-03 (Other: UNITE4TB under Innovative Medicines Initiative (IMI))
Record Dates: First submitted 2024-11-27; First posted 2024-12-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis
Keywords: Alpibectir; Ethionamide; Rifampicin; Pyrazinamide; Ethambutol; Adults; Newly Diagnosed; Drug- Susceptible; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Ethionamide; Isoniazid; Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 Arm 1 (A45E125) (Experimental): Alpibectir 45 mg once daily (OD) plus Ethionamide 125 mg OD
  Interventions: Drug: Alpibectir 45 mg once daily (OD) plus Ethionamide 125 mg OD
- Cohort 1 Arm 2 (A45E250) (Experimental): Alpibectir 45 mg OD plus Ethionamide 250 mg OD
  Interventions: Drug: Alpibectir 45 mg OD plus Ethionamide 250 mg OD
- Cohort 1 Arm 3 (HRZE) (Active Comparator): Isoniazid, rifampicin, pyrazinamide and ethambutol fixed dose combination, weight based
  Interventions: Drug: Isoniazid, rifampicin, pyrazinamide and ethambutol fixed dose combination, weight based
- Cohort 2 Arm 3 (HRZE) (Active Comparator): Isoniazid, rifampicin, pyrazinamide and ethambutol fixed dose combination, weight based
  Interventions: Drug: Isoniazid, rifampicin, pyrazinamide and ethambutol fixed dose combination, weight based
- Cohort 2 Arm 4 (A45E250RZE) (Experimental): Alpibectir 45 mg OD plus Ethionamide 250 mg OD plus Rifampicin 10 mg/kg OD plus Ethambutol 20 mg/kg OD plus Pyrazinamide 25 mg/kg OD
  Interventions: Drug: Alpibectir 45 mg OD plus Ethionamide 250 mg OD plus Rifampicin 10 mg/kg OD plus Ethambutol 20 mg/kg OD plus Pyrazinamide 25 mg/kg OD

INTERVENTIONS:
Drug: Alpibectir 45 mg once daily (OD) plus Ethionamide 125 mg OD — Cohort 1 Arm 1
  Arms: Cohort 1 Arm 1 (A45E125)
Drug: Alpibectir 45 mg OD plus Ethionamide 250 mg OD — Cohort 1 Arm 2
  Arms: Cohort 1 Arm 2 (A45E250)
Drug: Isoniazid, rifampicin, pyrazinamide and ethambutol fixed dose combination, weight based — Active Comparator
  Arms: Cohort 1 Arm 3 (HRZE); Cohort 2 Arm 3 (HRZE)
Drug: Alpibectir 45 mg OD plus Ethionamide 250 mg OD plus Rifampicin 10 mg/kg OD plus Ethambutol 20 mg/kg OD plus Pyrazinamide 25 mg/kg OD — Cohort 2 Arm 4
  Arms: Cohort 2 Arm 4 (A45E250RZE)

SUMMARY:
A multi-centre, randomized, open-label clinical trial. All treatments will be administered orally (PO) on days 1-14.

15 participants will be recruited into each treatment arm in two sequential cohorts. Each cohort will have participants enrolled onto the experimental regimen(s) or the standard of care (SOC; HRZE) control arm.

• Cohort 1 aims to generate safety data for a higher dose of alpibectir plus ethionamide 125 mg and 250 mg (arm 1: A45E125 and arm2: A45E250).

Once 5 participants have enrolled into arms 1 and 2 each, and completed 14 days of treatment, an interim safety review will be conducted to determine whether the study can advance to cohort 2.

• Cohort 2 will investigate safety of alpibectir and ethionamide (A45E250) in combination with rifampicin, pyrazinamide and ethambutol (A45E250RZE).

Participants on HRZE will serve as control for the EBA quantitative mycobacteriology in each cohort, and additionally as a safety benchmark for the A45E250RZE arm. The study is not statistically powered to make between arm comparisons of activity or safety. The treatment will not be blinded but the mycobacteriology laboratory staff performing the endpoint assays will remain blinded until analysis of the EBA results.

DETAILED DESCRIPTION:
This trial is designed to evaluate the antimycobacterial ejects and the safety of alpibectir in combination with other antimycobacterial agents, particularly Eto, over a 14-day period. The overarching objective is to optimise the dose of both alpibectir and ethionamide and to confirm the safety of the A45E250RZE regimen for future evaluation as an alternative regimen for INH mono-resistant TB. The data from the TASK-010 phase 2A and the ENABLE study will support evaluation of the optimal dose combination of AlpE to move forward into later phase studies. EBAs have historically been conducted between 2 and 14 days. This study will be a standard 14-day EBA design with multiple parallel and sequential treatment arms.

Cohort 1:

Arm 1 and 2: This cohort will add to the evidence base generated in the TASK-010 study (NCT05473195) to support dose optimisation of alpibectir and ethionamide (AlpE) and establish the safety of alpibectir 45 mg in humans, a dose which to date has not been evaluated.

Interim safety review: once a safety review of a subset of participants in arms 1 and 2 receiving the 45 mg dose of alpibectir is complete, cohort 2 will be permitted to begin recruiting once cohort 1 is complete.

Cohort 2:

Arm 4: will combine AlpE at doses determined to be safe and well tolerated from arms 1 and 2, with standard doses of rifampicin, isoniazid and ethambutol (A45E250RZE). Here AlpE replaces isoniazid in the regimen as part of the planned future use of the combination. This will establish the safety of this 5-drug combination at standard rifampicin doses. A well tolerated, adorable, oral, once daily dosing regimen would make the AlpE combination tolerable for patients and hence for the majority of people suffering from TB in less affluent regions of the world. All participants will remain under medical attention, and will be housed, and monitored in hospital from admission through day 15 of the treatment period; this will allow for continuous monitoring of the health status of each participant while initiating treatment, any of whom can be withdrawn at any stage of the trial and removed from study treatment should his/her condition suggest to the investigator that this would be in his/her best interest.

Biomarkers The traditional 2A proof-of-concept studies for new TB drugs also allow the exploration of new ways of measuring TB treatment activity in short-course trials beyond measurement of CFU or TTP. Each chemotherapeutic agent has the potential to contribute an interactive, often synergistic, role with other agents in a combination regimen, but this attribute is not captured by measuring decline in sputum CFU or TTP alone. Novel sputum biomarkers, and biomarkers from blood samples may have the potential to substitute or complement traditional sputum culture based methods to assess treatment responses. Host derived markers may also be able to describe the EBA of novel drugs.

Whole blood biomarkers:

Whole blood RNA analysis is emerging as a promising tool for the pathogen-free diagnosis and monitoring of TB treatment. This approach has the potential to revolutionize TB management by oqering a precise, individualized method to determine the duration of anti-TB therapy needed to achieve a relapse-free cure. The identification and validation of a 22-gene transcriptomic signature model (TB22) by Heyckendorf and colleagues serve as a significant advancement in this field. TB22 has shown superior performance in predicting individual treatment endpoints compared to 17 other publicly available RNA signatures. Specifically, TB22 demonstrated high accuracy in identifying end-of-therapy time points, with an AUC of 0.94 for predicting clinical outcomes. The model also indicated that cure could be achieved with significantly shorter treatment durations for patients with multidrug-resistant TB (MDR-TB). Whole blood will be collected in participants who consent for evaluation of whole blood RNA in models like the TB22 or others investigating the use of novel biomarkers.

Sputum biomarkers:

The Molecular Bacterial Load Assay (TB-MBLA) and PATHFAST (LAM) are novel biomarkers being evaluated for their potential to improve TB treatment monitoring. The TB-MBLA oqers a rapid and precise measurement of bacterial load by detecting RNA, which is less aqected by the presence of non-culturable bacteria. This assay, coupled with appropriate RNA preservatives, can provide real-time insights into the bacterial burden and treatment eqicacy. PATHFAST (LAM) focuses on detecting lipoarabinomannan (LAM) in sputum, a component of the mycobacterial cell wall. LAM detection can serve as a biomarker for active TB, providing an additional layer of diagnostic information. Its integration into treatment monitoring can help assess the eqicacy of TB drugs, particularly in reducing bacterial load in the lungs. These biomarkers will be evaluated for use as secondary and exploratory endpoints in 2A setting within this protocol.

Study Drug Rationale Given the increasing need for novel regimens and highly eqective, well-tolerated drugs to treat participants with TB, it is important to evaluate the antituberculosis activity of established anti- TB drugs that have been enhanced to generate higher eqicacy, lower adverse eqects, or both. These evaluations should occur in a carefully conducted, controlled, and standardised EBA study to determine their contributions as building blocks for potential future studies of new regimens. The results of this study will be used to support future studies of longer duration. Activity rationale: Extending the EBA duration from 7 to 14 days is informed by data suggesting that the full antimycobacterial eqect of alpibectir may not be completely observable within the 7-day period, thus a longer duration allows for a more accurate assessment of its activity and safety. The absence of human data at this dose level warrants careful monitoring, but the potential benefits of a more eqective treatment regimen for INH-resistant and other DR-TB justify this exploration. Safety rationale: The inclusion of a 45 mg dose of alpibectir in this study, despite not having been tested in previous phase 1 or 2 trials, is expected to be safe and well tolerated. Appropriate safety measures are in place to monitor participants throughout their treatment and evaluation of this premise. Pharmacodynamic scaling from pre-clinical models to humans suggests that the higher dose is likely to maximize therapeutic activity while maintaining a favourable safety profile. Given the promising preclinical and phase 2A results, it is both scientifically justified and ethically responsible to optimise the dose of alpibectir in a controlled clinical trial. The trial design includes comprehensive safety assessments to identify and manage any adverse events promptly. The investigation of 14 days in a 5-drug regimen (A45E250RZE) will provide crucial pilot safety and tolerability data. Hepatotoxic eqects associated with RZE-based regimens may occur later in treatment, and therefore 14-day data will provide some evidence on the safety of the regimen when moving into later phases of development. This approach ensures that any potential hepatotoxic eqects or other adverse events are identified and managed early, thereby safeguarding participants and informing future phase studies.

Control rationale: HRZE is being used as the control arm as the current SOC for PTB. Using HRZE allows for a direct comparison of the safety of the diqerent study arms against WHO approved regimen, and a microbiological control.

Rationale for the Selection of the Agents and Doses Alpibectir Alpibectir increases intra-bacterial bioactivation of Eto and as such works in combination with Eto to enhance Eto exposure in TB without increasing the dose of Eto. The selection of a 45 mg dose of alpibectir is based on pharmacodynamic scaling from animal models to humans, which indicates that this dose is likely to maximize therapeutic activity while maintaining a favourable safety profile, as evidenced by substantial bacterial load reduction in preclinical trials. Preclinical data showing that alpibectir at doses of up to 1.6 mg/kg prevented mortality in a BALB/c mouse model, suggesting a protective eqect of the drug at higher doses. Combination therapy arms with alpibectir and Eto are grounded in the compound's ability to enhance the bactericidal effect of Eto, as proven in pre-clinical trials and the recent phase 2 EBA. The trial seeks to further evaluate the potential of reducing the effective dose of Eto required, thus potentially reducing the drug's side effects, and enhancing patient tolerability.

Regimens explored in the TASK-010 trial evaluating doses of 9 mg and 27 mg of alpibectir along with Eto 120-500 mg, when pooled with the ENABLE 45 mg alpibectir and 125-250 mg Eto will support PKPD modelling and establish a robust dose-response curve to support the best dose combination.

Ethionamide Two doses of Eto will be used in this study, 125 mg, and 250 mg. EBA was seen in both doses when combined with alpibectir 27 mg in the recent TASK-010 phase 2a trial, these doses were also well tolerated in participants. The aim is to maintain a low, active dose of Eto in combination with alpibectir to ensure tolerability.

Rifampicin (A45E250RZE) The inclusion of a combination arm with alpibectir, Eto and RZE (Rifampicin, Pyrazinamide and Ethambutol) is designed to evaluate the EBA of the combination as part of a comprehensive TB treatment regimen. This could potentially inform the design of further trials. Additionally, we aim to assess whether the AlpE combination can serve as a viable alternative INH, particularly in situations where INH cannot be used due to resistance or other contraindications. This study will focus on the safety of the A45E250RZE combination.

Pyridoxine All participants will receive pyridoxine as prophylaxis against isoniazid-related or ethionamide related peripheral neuropathy, as per the National TB Guidelines. Currently this is 25 mg orally once daily, or with each dose of isoniazid or ethionamide.

ART Using the multi-cohort design, the early safety of the AlpE combination at higher alpibectir doses will be determined, as well as the safety of the A45E250RZE combination. In South Africa, between 1/3 and ½ patients diagnosed with TB are co-infected with HIV. It is important to understand the impact ART will have on the activity of any TB drug or regimen. As such, we have elected to include participants with HIV/TB co-infection who are receiving one of a limited number of ART options currently recommended as first line therapy. Inclusion of this critical group is unlikely to have significant impact either on the activity of the regimens, or on the efficacy of the ART as determined by the known effect of each drug on inhibiting or inducing various substrates involved in metabolism. This allows the study to generate early safety data with minimal risk to the participants. The ART regimens permitted include 2 non-nucleoside reverse transcriptase inhibitors (NRTI) and dolutegravir. The NRTI's permitted may include Emtricitabine, Lamivudine and/or Tenofovir.

Dolutegravir (Mondleki, 2022):

* Dolutegravir does not induce or inhibit metabolising enzymes. Dolutegravir is a substrate of the drug efflux pumps P-gp and BCRP. It is primarily metabolised by enzyme UGT1A1, and to a smaller degree by CYP3A4, and UGT1A3 and 1A9.
* Alpibectir has a minimal risk of inhibition of CYP3A4, P-gp, and BCRP (section 3.1). No information is available about the effect of alpibectir on UGT1A1, although in vitro work is planned and will be conducted. INH has a small effect on CYP3A4 inhibition, this effect may be more pronounced in slow acetylators though the clinical effect is likely modest.
* Based on the currently available data in which lower concentrations of dolutegravir were found when co-administered with rifampicin but not impact on viral suppression was demonstrated, a clinically significant drug-drug interaction between dolutegravir and the AlpE combination or HRZE are not anticipated (Sekaggya-Wiltshire, 2023). Current South African Department of Health guidelines recommend increasing the dose of dolutegravir to 50 mg twice daily (from 50 mg daily)(Primary Care Guide, 2021). This will be implemented in participants randomized to arms receiving rifampicin.

Emtricitabine, Lamivudine, Tenofovir (NRTIs)

* Emtricitabine, lamivudine and tenofovir are not substrates or inhibitors of CYP enzymes but are substrates for various transporter proteins. For example, Tenofovir is a substrate of BCRP/ABCG2 and P-glycoprotein/ABCB1, and an inhibitor of MRP2 (Wassner, 2020).
* Based on the currently available data, a clinically significant drug-drug interaction between the NRTIs and the AlpE combination or RZE are not anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures and willing to adhere to all required study procedures and restrictions for the duration of the trial.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed and untreated for this episode of pulmonary TB.
5. Rifampicin- and isoniazid susceptible pulmonary TB as determined by molecular testing (GeneXpert XDR or Genotype MTBDRplus for INH).
6. A chest X-ray taken during the screening period or up to 2 weeks before screening which, in the opinion of the investigator, is consistent with TB.
7. GeneXpert positive with a quantitative readout of medium or high.
8. Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 ml or more).
9. Be of non-childbearing potential or of childbearing potential using effective methods of birth control, as defined in section 5.2 and in Appendix 1.

   Female Participants
10. For WOCBP who are not already receiving contraception per Appendix 1 requirements, agree to receive injectable or other contraceptive methods (per Appendix 1), to be given during screening, and at least 1 day prior to first dose of IMP.

    Male Participants
11. Agree to ALL of the following during the study intervention period and for at least 90 days, after the last dose of study intervention:

    1. Refrain from donating fresh unwashed semen
    2. Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.

Exclusion Criteria:

1. Evidence of clinically significant conditions or findings, other than TB, that might compromise safety or the interpretation of trial endpoints, per discretion of the investigator.
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the investigator.
3. History of epilepsy, seizures or other neuropsychiatric disorders that might compromise safety or the interpretation of trial endpoints, per discretion of the investigator.
4. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, persistent jaundice (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. History of hypothyroidism
6. QTcF of >450 ms at baseline
7. Clinically significant evidence of extra-thoracic TB, as judged by the investigator.
8. History of allergy to any of the trial IMP as confirmed by the clinical judgement of the investigator.
9. Alcohol or drug abuse, that in the opinion of the investigator, is sufficient to compromise the safety or cooperation of the participant.
10. HIV positive AND:

    1. CD4 < 250cells/mm3
    2. On other ART regimen not listed below or, if not on ART they are not willing to wait to start treatment until completion of study regimen

    Note: ART regimens permitted is limited to the following in line with local guidelines for 1st line ART:
    * NRTIs selected from: Emtricitabine, Lamivudine, Tenofovir
    * PLUS Dolutegravir 50 mg daily, or 50 mg twice daily if randomized to a rifampicin containing arm.

    Participants established on ART (2 NRTIs and dolutegravir) for more than 30 days at start of screening are eligible for participation.

    As the drug-drug interaction potential of ART has not been fully investigated with the IMP, NNRTIs (efavirenz, nevirapine) and other protease inhibitors will not be permitted in this study.
11. Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of trial participation and for at least 90 days after the last dose of study intervention. Male participant planning to conceive a child for at least 90 days, after the last dose of study intervention in the trial.

    Treatment History
12. Participation in other clinical studies with investigational agents within 8 weeks prior to screening.
13. Treatment received for this episode of TB with any drug active against M. tb (including but not limited to isoniazid, ethambutol, cycloserine, fluoroquinolones, rifamycins, aminoglycosides, nitroimidazoles, bedaquiline, oxazolidinones, para-amino salicylic acid, pyrazinamide, thioacetazone, thioamides).
14. Treatment with immunosuppressive medications such as TNF-alpha inhibitors within 2 weeks prior to screening, or systemic corticosteroids for more than 7 days within 2 weeks prior to screening.
15. Unavoidable treatment with prohibited concomitant medications (see section 5.3.2) anticipated during administration of IMP.

    Laboratory Safety Testing
16. Presence of hepatitis B surface antigen (HBsAg+)
17. Positive hepatitis C antibody test result (HCV IgG+)
18. Participants with the following toxicities at screening as defined by the enhanced CTCAE toxicity table:

    1. creatinine >1.5 times upper limit of normal (ULN)
    2. haemoglobin <8.0 g/dL
    3. platelets <50x109 cells/L
    4. serum potassium <3.0 mmol/L
    5. alanine aminotransferase (ALT) ≥5 x ULN
    6. total bilirubin >1.5 x ULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5 x ULN as long as direct bilirubin is ≤1.5xULN
    7. Total white cell count <1.5 cells/L
    8. Thyroid Stimulating Hormone > ULN
    9. Glucose < 3.5 mmol/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
EBA-TTP (0-14) | 14 days
  The EBA TTP (0-14) as determined by the rate of change in log10TTP in sputum over the period day 0 (baseline sample) to Day 14 will be described using linear, bi-linear, or non-linear functions using nonlinear mixed effects modelling of log10TTP over time. Estimates of rates of change including uncertainties for each treatment group will be given and graphically illustrated.

SECONDARY OUTCOMES:
EBA CFU (0-14) | 14 days
  The EBA CFU (0-14) as determined by the rate of change in log10CFU per ml sputum over the period day 0 to day 14 will be described using linear, bi-linear, or non-linear functions using nonlinear mixed effects modelling as dictated by the data of log10CFU over time. Estimates of rates of change including uncertainties for each treatment group will be given and graphically illustrated.
EBA (0-2) and EBA (2-14) | 2-14 days
  The EBA (0-2) and EBA (2-14) determined by the rate of change in The EBA (0-2) and EBA (2-14) determined by the rate of change in log10CFU and log10TTP over time.
Safety and tolerability | 14 days
  The incidence of the following events will be summarized by treatment group:
  * Incidence of treatment-emergent adverse events (TEAEs).
  * Incidence of TEAEs by Severity.
  * Incidence of drug related TEAEs.
  * Incidence of Serious TEAEs.
  * Incidence of TEAEs leading to treatment discontinuation.
  * Incidence of TEAEs leading to early withdrawal from the study.
  * Incidence of TEAEs leading to death. Descriptive summary statistics will be presented for other safety variables: laboratory parameters, physical examination, vital signs, concomitant medication
PK analysis - Cmax | 14 days
  Maximum observed plasma drug concentration (Cmax),
Biomarkers (Sputum) | 14 days
  The EBA MBLA (0-14) and EBA LAM (0- 14) as determined by the rate of change in biomarker over the period day 0 to day 14 will be described using linear, bi-linear, or non-linear functions using nonlinear mixed effects modelling as dictated by the data of biomarker over time. Estimate of rates of change including uncertainties for each treatment groups will be given and graphically illustrated. treatment arm, based on the mycobacterial load assay (MBLA) and PATHFAST TB Lipoarabinomannan (LAM) test.
Biomarkers (Whole Blood) | 14 days
  Descriptive statistics will be computed for each biomarker.
Mycobacterial parameters | 2-14 days
  Cultures from baseline (Day -2, Day -
  1) and post-baseline (Day 14) will be kept. In case end of treatment cultures are not available the last available culture after day 8 will be kept. Determination of the minimum inhibitory concentration (MIC) of the investigational agents will be done. If a significant MIC shift (≥4-fold) of these drugs is observed, MIC determination of all regimen agents will be triggered and genome sequencing of isolates with the shift in MIC will be performed.
Drug-drug interaction - AUC (0-24) | 14 days
  The AUC (0-24) of alpibectir with and without rifampicin will be compared.
PK Analysis (AUC (0-24), AUC (0-∞), AUC(0-tau) | 14 days
  Area under the plasma drug concentration versus time curve ((AUC (0-24), AUC (0-∞), AUC(0-tau))
PK Analysis (Tmax) | 14 days
  Time to maximum observed plasma drug concentration (Tmax),
PK Analysis - apparent terminal half-life (t1/2) | 14 days
  Apparent terminal half-life (t1/2), as appropriate will be estimated for alpibectir, Eto and Eto-SO using a noncompartmental approach.
PK Analysis-Descriptive Statistics | 14 days
  Mean, standard deviation, coefficient of variation, median, minimum, and maximum, geometric mean, and geometric mean coefficient of variation (CV)% will be computed for each PK parameter.
Drug-drug interaction - Cmax | 14 days
  The Cmax of alpibectir with and without rifampicin will be compared.
Drug-drug interaction - Tmax | 14 days
  The Tmax of alpibectir with and without rifampicin will be compared.
  [

CONTACTS AND LOCATIONS:
Overall Officials: Gifty Okyere-Manu, MBChB, Principal Investigator — TASK
Locations (1):
- TASK, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
Data will be shared based on the following principles:
  No data should be released that would compromise an ongoing trial or study. There must be a strong scientific or other legitimate rationale for the data to be used for the requested purpose. Investigators who have invested time and effort into developing a trial or study should have a period of exclusivity in which to pursue their aims with the data, before key trial data are made available to other researchers. The resources required to process requests should not be under-estimated, particularly successful requests which lead to preparing data for release. Therefore adequate resources must be available in order to comply in a timely manner or at all, and the scientific aims of the study must justify the use of such resources. Data exchange complies with Information Governance and Data Security Policies in all of the relevant countries.

REFERENCES:
- See also: SANCTR — https://sanctr.samrc.ac.za/Admin/Home.aspx